CLINICAL TRIAL: NCT03994289
Title: Effects of Motor-assisted Cycling and Functional Electrical Stimulation Cycling on Postprandial Glucose in Type 2 Diabetic Patients With Activities of Daily Living Disability
Brief Title: Motor-assisted Cycling and FES Cycling for Postprandial Glucose in Diabetic Patients With ADL Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Chong Lee, Associate Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00008262
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Type2 Diabetes; Disability Physical
Keywords: exercise; FES
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants remain seated for 2 hours after the intake of a standardized breakfast.
- Motor-assisted cycling (Experimental): Participants will perform 3 bouts of motor-assisted cycling, each bout lasting 10 minutes, after the intake of a standardized breakfast.
  Interventions: Behavioral: Motor-assisted cycling
- FES cycling (Experimental): Participants will perform 3 bouts of FES cycling, each bout lasting 10 minutes, after the intake of a standardized breakfast.
  Interventions: Behavioral: FES cycling

INTERVENTIONS:
Behavioral: Motor-assisted cycling — Participants will perform the motor-assisted cycling exercise using a physical therapy bike (RECK; Betzenweiler, Germany). Participants will perform 3×10-min bouts of motor-assisted cycling at the highest tolerable cadence. Before each bout, participants will perform 1-2 minutes of motor-assisted cycling at 5-10 rpm as a warm-up.
  Arms: Motor-assisted cycling
Behavioral: FES cycling — The testing procedures will be identical to that in the motor-assisted cycling visit except for the exercise type. Participants will wear FES cuffs on the upper and lower legs, bilaterally.
  . The FES cycling will be performed on the motor-assisted bike using the wearable FES equipment. The purpose of motor-assisted cycling is to provide constant cadence. The Bioness L300 Plus system (Bioness, Valencia, CA) will be worn on the upper and lower legs to stimulates the quadriceps and dorsiflexors muscles during the motor-driven cycling exercise. An embedded gyroscope of the cuff can detect the motion of the lower leg so that the electrical stimulations will be generated at appropriate timing to activate leg muscles during the cycling exercise.
  Arms: FES cycling

SUMMARY:
Exercise has been the cornerstone of diabetes management. However, many diabetic patients have ADL disabilities and experience substantial difficulty in performing usual exercises, such as brisk walking and upright cycling. There is an urgent need to provide alternative exercise modalities for diabetic patients with ADL disabilities. In this study, investigators will investigate the effects on the glucose of three exercise modalities, including motor-assisted cycling (i.e., cycling on a motor-driven bike) and functional electrical stimulation (FES) cycling, during which the investigators will use electrical current to facilitate cycling movements.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years.
* Physician-diagnosed type 2 diabetes.
* ADL disability (self-reported).

Exclusion Criteria:

* Fasting glucose ≥ 250 mg/dL.
* Symptomatic hypoglycemic events in the past three months.
* Insulin injection or infusion
* Systolic blood pressure ≥ 160 mmHg OR Diastolic blood pressure ≥ 100 mmHg
* Diagnosis of NYHA class I-IV heart failure
* Myocardial infarction in the past 6 months
* Recent or current angina, shortness of breath, or other symptoms suggestive of heart failure
* Diagnosed Cancer
* Unable to consent due to impaired cognitive function
* Bone fracture, joint dislocation, or joint stiffness
* Local skin disorders at the FES cuff area or CGM sensor area
* Implantable electronic or metallic devices, such as cardioverter defibrillator and pacemaker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose AUC | The glucose will be measured using CGM during the 2-hour postprandial period.

CONTACTS AND LOCATIONS:
Locations (1):
- Brookdale Senior Living Central Chandler, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: No